CLINICAL TRIAL: NCT07366359
Title: Comparison of the Effectiveness of Labor Induction Using Dinoprostone Followed by Oxytocin Versus Oxytocin Alone in Term Pregnancies With Premature Rupture of Membranes and an Unfavorable Cervix - A Randomized Clinical Trial
Brief Title: PGE2 Followed by Oxytocin vs Oxytocin in Term PROM (POXY-PROM)
Acronym: POXY-PROM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Hospital of Obstetrics and Gynecology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHOG.2025.POXY-PROM
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Premature Rupture of Fetal Membranes; Labor, Induced; Cervical Ripening
Keywords: Premature Rupture of Fetal Membranes; Labor Induction; Dinoprostone; Oxytocin; Cervical Ripening; Vaginal Delivery
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Dinoprostone; Oxytocin

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel study arms: (1) cervical ripening with a 6-hour vaginal dinoprostone insert (Propess) followed by oxytocin if needed, or (2) immediate induction with intravenous oxytocin. All participants remain in their assigned arm throughout the study; no crossover occurs. Randomization is computer-generated and allocation is concealed. Both interventions reflect routine clinical practice for term PROM with an unfavorable cervix.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dinoprostone (Propess) + Oxytocin (Experimental): Participants in this arm will receive a 10-mg vaginal dinoprostone insert (Propess) for cervical ripening. After 6 hours, if active labor has not begun or uterine contractions are inadequate, intravenous oxytocin will be started according to the hospital's standardized induction protocol. Continuous fetal monitoring and standardized management of uterine tachysystole will be applied. This approach reflects a sequential induction method commonly used for women with term PROM and an unfavorable cervix.
  Interventions: Drug: Sequential Induction: Dinoprostone Followed by Oxytocin
- Immediate Oxytocin Induction (Active Comparator): Participants in this arm will receive immediate induction of labor using intravenous oxytocin according to the hospital's standardized induction protocol. No cervical ripening agent will be used before starting oxytocin. Maternal and fetal status will be monitored throughout labor, and uterine tachysystole will be managed in line with institutional guidelines. This arm represents the comparator strategy of inducing labor directly with oxytocin in women with term PROM and an unfavorable cervix.
  Interventions: Drug: Immediate Oxytocin Induction

INTERVENTIONS:
Drug: Sequential Induction: Dinoprostone Followed by Oxytocin — A sequential induction strategy in which a 10-mg vaginal dinoprostone insert (Propess) is placed for cervical ripening. After 6 hours, if active labor has not begun or uterine contractions are inadequate, intravenous oxytocin is initiated according to the hospital's standardized induction protocol. Continuous fetal monitoring is applied, and tachysystole is managed per institutional guidelines.
  Other Names: Dinoprostone (Propess)
  Arms: Dinoprostone (Propess) + Oxytocin
Drug: Immediate Oxytocin Induction — Intravenous oxytocin is used for immediate induction of labor in women with term prelabor rupture of membranes and an unfavorable cervix. Oxytocin is started according to the hospital's standardized induction protocol without prior use of cervical ripening agents. Maternal and fetal status are monitored throughout labor, and uterine tachysystole is managed according to institutional guidelines.
  Other Names: Oxytocin
  Arms: Immediate Oxytocin Induction

SUMMARY:
This study is being done to learn more about the best way to start labor for pregnant women whose water breaks at term before labor begins, a condition called term prelabor rupture of membranes (term PROM). When this happens and the cervix is not ready for labor, it is unclear which induction method works best and is safest for mother and baby.

The purpose of this study is to compare two common ways to induce labor in women with term PROM and an unfavorable cervix (Bishop score ≤ 6). One group will receive a vaginal dinoprostone insert (Propess) for 6 hours to soften the cervix, followed by oxytocin if labor does not start. The other group will receive immediate oxytocin through a vein.

Pregnant women aged 18 years or older with a single baby in head-down position at 37-42 weeks, whose water has broken and whose cervix is not yet favorable, may be able to join this study. All care will be provided at the National Hospital of Obstetrics and Gynecology in Hanoi, Vietnam, where both medicines are already used in routine practice.

The main outcome is how many women have a vaginal birth. The study will also look at how long it takes from induction to birth, complications for mothers and babies, and women's experiences of labor. The results may help doctors choose the safest and most effective way to induce labor for women with term PROM in the future.

DETAILED DESCRIPTION:
Prelabor rupture of membranes at term (term PROM) occurs in approximately 8% of pregnancies and is associated with increased risks of maternal infection, neonatal morbidity, and cesarean delivery when labor does not begin promptly. International guidelines recommend active induction of labor for women with term PROM; however, the optimal induction strategy for women presenting with an unfavorable cervix (Bishop score ≤ 6) remains uncertain.

Oxytocin is widely used for induction of labor and is effective when the cervix is favorable, but its efficacy may be reduced in the presence of an unripe cervix. Prostaglandin E2 (dinoprostone) is commonly used for cervical ripening and may improve the likelihood of vaginal delivery when administered prior to oxytocin. Previous randomized trials comparing dinoprostone followed by oxytocin with oxytocin alone have suggested potential benefits, but the available evidence is limited by small sample sizes and inconsistent results. Additional high-quality randomized evidence is therefore required to guide clinical practice in this population.

This randomized controlled trial compares two induction strategies for women with term PROM and an unfavorable cervix: (1) cervical ripening using a 6-hour vaginal dinoprostone (Propess) insert followed by intravenous oxytocin if labor has not commenced, and (2) immediate induction with intravenous oxytocin alone. Both interventions are routinely used in clinical practice in Vietnam and are considered safe.

Participants are randomly assigned in a 1:1 ratio using a computer-generated randomization sequence with variable block sizes of 4 and 6, with allocation concealment ensured through centralized randomization. Randomization is performed after confirmation of eligibility and completion of the informed consent process. Participants remain in their assigned study arm throughout the trial, and no crossover between arms is permitted. All aspects of intrapartum care, including fetal heart rate monitoring, assessment of labor progress, and management of uterine tachysystole or other complications, are conducted according to standard institutional protocols.

The primary outcome of the study is vaginal delivery. Secondary outcomes are selected in accordance with the internationally developed core outcome set for trials on induction of labour and include key maternal, neonatal, and patient-reported outcomes. Maternal outcomes include mode of delivery, time from induction to delivery, need for oxytocin augmentation, uterine hyperstimulation, postpartum hemorrhage, maternal infection, admission to intensive care, hysterectomy, and maternal death. Neonatal outcomes include Apgar scores, admission to the neonatal intensive care unit, neonatal infection, hypoxic-ischemic encephalopathy or need for therapeutic hypothermia, and neonatal death. Patient-reported outcomes, including overall labor pain and maternal satisfaction with the birth process, are also assessed.

A total sample size of 450 participants has been calculated to provide adequate statistical power while accounting for potential attrition. The findings of this study are expected to clarify whether cervical ripening with dinoprostone prior to oxytocin induction improves clinically meaningful outcomes for women with term PROM and an unfavorable cervix, and may help inform future national and international guidelines on induction of labor.

ELIGIBILITY:
Inclusion Criteria

* Maternal age ≥ 18 years
* Gestational age from 37 to 42 weeks, determined by last menstrual period or by a first- or second-trimester ultrasound
* Live singleton fetus
* Prelabor rupture of membranes (PROM) confirmed by at least one of the following:

  * Amniotic fluid visibly draining from the cervical os during sterile speculum examination
  * Pool of fluid in the posterior fornix
* Cephalic presentation
* Bishop score ≤ 6
* No spontaneous uterine contractions
* No contraindications for vaginal delivery

Exclusion Criteria:

* Active labor
* Previous uterine surgery (e.g., cesarean section)
* Chorioamnionitis or non-reassuring fetal status
* Major fetal anomalies
* Contraindications to prostaglandin or vaginal delivery
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal delivery | From induction until delivery, assessed up to 36 hours after randomization
  Number of participants delivered vaginally

SECONDARY OUTCOMES:
Mode of delivery | Within 24 hours from labor induction
  Number of participants according to mode of delivery, categorized as vaginal delivery, operative vaginal delivery (forceps), or cesarean section
Time from induction of labor to delivery | From induction until delivery, assessed up to 24 hours after induction
  Duration from induction of labor to delivery (hours)
Oxytocin augmentation | From induction until delivery, assessed up to 24 hours after induction
  Number of participants in the intervention group (Group I) who received intravenous oxytocin during the induction process
Uterine hyperstimulation | From induction until delivery, assessed up to 24 hours after induction
  Number of participants who experienced uterine hyperstimulation, defined as more than 5 uterine contractions in 10 minutes over a minimal period of two consecutive 10-minute intervals, and/or a single uterine contraction lasting more than 3 minutes with fetal heart rate changes
Maternal satisfaction | Once between 90 minutes and 3 hours after delivery
  Maternal satisfaction, assessed using a 5-point Likert scale, where 1 indicates very dissatisfied and 5 indicates very satisfied
Haemorrhage | Within 24 hours from delivery
  Number of participants who experienced postpartum haemorrhage, defined as estimated blood loss greater than 500 mL after vaginal birth or greater than 1000 mL after caesarean birth within 24 hours after delivery
Uterine rupture | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants with uterine rupture
Hysterectomy for any complications resulting from birth | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants who underwent hysterectomy for any complication resulting from childbirth
Maternal infection | From induction until maternal hospital discharge, assessed up to 28 days after induction
  Number of participants with maternal infection, defined as the presence of at least one of the following criterias:
  Fever (defined as a temperature ≥38.0 degrees Celsius). Start of intravenous broad-spectrum antibiotics (with evidence of infection confirmed by clinical and subclinical presentation).
  Endometritis, myometritis or urinary tract infection (proven positive vaginal discharge/urine culture).
Damage to internal organs | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants with injury to internal organs, including intestines, bladder, or ureters, diagnosed clinically and/or confirmed intraoperatively during delivery or postpartum care.
Intensive care admission | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants admitted to the intensive care unit
Cardiorespiratory arrest | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants who experienced cardiorespiratory arrest
Pulmonary embolus | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants diagnosed with pulmonary embolism
Stroke | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants diagnosed with stroke
Maternal death | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants who died from any cause between randomization and maternal hospital discharge
Length of maternal hospital stay | From admission until maternal hospital discharge, assessed up to 28 days after admission
  Duration of stay in hospital (days)
Birth trauma | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates with birth trauma, defined as the presence of at least one birth-related traumatic injury, including bone fracture, traumatic pneumothorax, facial nerve palsy, brachial plexus injury, or other clinically diagnosed birth-related trauma, identified by clinical examination and/or imaging during the neonatal hospital stay
Hypoxic ischaemic encephalopathy or need for therapeutic hypothermia | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates with hypoxic ischemic encephalopathy or need for therapeutic hypothermia
Meconium aspiration syndrome | From delivery until neonatal hospital discharge, assessed up to 07 days after delivery
  Number of neonates diagnosed with meconium aspiration syndrome, defined by the presence of:
  Meconium-stained amniotic fluid Respiratory distress at birth or shortly after birth Characteristic radiographic features: The initial chest film may show streaky, linear densities -> the lungs typically appear hyper-inflated with flattening of the diaphragms.
Need for respiratory support | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates requiring respiratory support, defined as the use of one or more of the following interventions within the first 72 hours after birth: Endotracheal intubation; Continuous Positive Airway Pressure (CPAP); High-flow nasal cannula (HFNC); Use of respiratory support as part of ventilation or cardiopulmonary resuscitation.
Neonatal infection | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates diagnosed with neonatal infection, defined as meeting at least one of the following criteria:
  Presence of a clinically ill neonate in whom systemic infection is suspected and confirmed by a positive blood culture, cerebrospinal fluid (CSF) culture, or catheterized/suprapubic urine culture; Or, in the absence of positive cultures, clinical evidence of cardiovascular collapse consistent with infection; Or radiographic evidence (e.g., chest X-ray) confirming infection.
Neonatal seizures | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates with neonatal seizures
Neonatal death | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates who died during the intrapartum period, neonatal period, or perinatal period
Admission to the neonatal unit | From delivery until neonatal admission, assessed up to 7 days after delivery
  Number of neonates admitted to the neonatal unit

OTHER OUTCOMES:
Vaginal delivery within 12 hours | From induction until delivery, assessed up to 12 hours after induction
  Number of participants delivered vaginally within 12 hours
Reaching active phase of labor | From induction until reaching active phase, assessed up to 12 hours after induction
  Number of participants who developed regular uterine contractions accompanied by cervical dilation of ≥5 cm, as assessed by a qualified obstetric provider
Time from induction to dinoprostone insert removal | From induction until dinoprostone vaginal insert removal, assessed up to 12 hours after induction
  Duration from induction to dinoprostone vaginal insert removal (hours). Applicable to participants in the dinoprostone insert arm only
Time from induction to active phase of labor | From induction until reaching active phase of labor, assessed up to 12 hours after induction
  Duration from induction to active phase of labor (hours)
Time from membrane rupture to induction | From membrane rupture until initiation of labor induction, assessed up to 24 hours after membrane rupture
  Duration from the first confirmed rupture of membranes (either by maternal report of clear fluid leakage or clinical diagnosis) to the initiation of labor induction (hours)
Time from membrane rupture to delivery | From membrane rupture until delivery, assessed up to 36 hours after membrane rupture
  Duration from the first confirmed rupture of membranes (either by maternal report of clear fluid leakage or clinical diagnosis) to delivery (hours).
Time from intrapartum antibiotic prophylaxis to delivery | From the first dose of intrapartum antibiotic prophylaxis until delivery
  Time interval (in hours) from the first dose of intravenous intrapartum antibiotic prophylaxis to delivery
Meconium-stained amniotic fluid | From membrane rupture until delivery, assessed up to 36 hours after membrane rupture
  Number of participants with meconium-stained amniotic fluid, defined as the presence of meconium in the amniotic fluid, as documented by clinical staff during labor or at delivery
Use of tocolysis for excessive uterine activity | From induction until delivery, assessed up to 24 hours after induction
  Number of participants who required tocolytic treatment due to excessive uterine activity during labor induction
Maternal side effects related to labor induction | From induction until delivery, assessed up to 24 hours after induction
  Number of participants experiencing maternal side effects related to labor induction, including nausea, vomiting, diarrhea, or other gastrointestinal symptoms
Use of analgesia during labor | From induction until delivery, assessed up to 24 hours after induction
  Number of participants who received any form of analgesia during labor, including epidural analgesia, systemic opioids (e.g., fentanyl), or other pharmacological pain relief methods
Postpartum blood transfusion | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants having maternal post-partum blood transfusion
Uterine atony | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants with uterine atony requiring treatment with two or more uterotonic agents other than oxytocin and/or additional interventions, including manual uterine compression, compression sutures, uterine artery ligation, embolization, hypogastric artery ligation, or balloon tamponade
Hysterectomy | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants who underwent hysterectomy for any postpartum complication
Group B Streptococcus colonization | From diagnosis to delivery
  Number of participants with Group B Streptococcus (GBS) colonization, defined as a positive screening test for Streptococcus agalactiae during the late third trimester
Overall labor pain | Assessed once between 90 minutes and 3 hours after delivery
  Maternal overall pain experienced during labor, assessed using a 0-10 Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable
Composite maternal outcome | From randomization until maternal hospital discharge, assessed up to 28 days after randomization
  Number of participants with at least one of the following maternal complications: chorioamnionitis, postpartum hemorrhage, intensive care unit admission, hysterectomy, uterine rupture, cervical tear, or maternal death
Apgar score at 1 minute | Assessed at 1 minute after birth
  Apgar score assessed at 1 minute after birth
Apgar score at 5-minute | Assessed at 5-minute after birth
  Apgar score assessed at 5-minute after birth
Low Apgar score at 1 or 5-minute | Assessed at 1 and 5-minute after birth
  Number of neonates with an Apgar score of 7 or less at 1 or 5-minute after birth
Admission to neonatal intensive care unit | From delivery until NICU admission, assessed up to 7 days after delivery
  Number of neonates admitted to the Neonatal Intensive Care Unit (NICU)
Reasons for NICU admission | From delivery until Neonatal Intensive Care Unit admission, assessed up to 28 days after delivery
  Reason for Neonatal Intensive Care Unit admission such as: respiratory distress, hypoglycemia, seizures, etc..
Length of NICU stay | From admission to Neonatal Intensive Care Unit until neonatal discharge or hospital referral, assessed up to 28 days after Neonatal Intensive Care Unit admission
  Duration from admission to Neonatal Intensive Care Unit to Neonatal Intensive Care Unit discharge or hospital referral
Neonatal hypoglycemia | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates with hypoglycemia
Neonatal jaundice and hyperbilirubinemia | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates diagnosed with jaundice and hyperbilirubinemia during the neonatal hospital stay
Intracranial hemorrhage | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery.who received blood transfusion
  Number of neonates diagnosed with intracranial hemorrhage, defined as any bleeding within the cranial vault confirmed by clinical assessment and/or imaging studies, including intraventricular hemorrhage, subdural hemorrhage, subarachnoid hemorrhage, or subgaleal hemorrhage
Neonatal blood transfusion | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates who received blood transfusion during the neonatal hospital stay
Neonatal hospital referral | From delivery until neonatal hospital referral, assessed up to 28 days after delivery
  Number of neonates referred to another hospital due to severe neonatal complications
Composite neonatal outcome | From delivery until neonatal hospital discharge, assessed up to 28 days after delivery
  Number of neonates experiencing at least one of the following events: low Apgar score, prematurity, neonatal intensive care unit admission, neonatal infection, neonatal seizures, respiratory distress syndrome, intraventricular hemorrhage, necrotizing enterocolitis, or perinatal death

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital of Obstetrics and Gynecology, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not yet decided whether individual participant data will be shared. As the study has not yet been conducted, there is currently limited information regarding the effectiveness of the interventions and potential risks. The decision on data sharing will depend on future considerations, including institutional policies, ethical approvals, and the establishment of appropriate data governance and data sharing agreements to ensure participant confidentiality.

REFERENCES:
- [Result] Prelabor Rupture of Membranes: ACOG Practice Bulletin, Number 217. Obstet Gynecol. 2020 Mar;135(3):e80-e97. doi: 10.1097/AOG.0000000000003700. PMID 32080050
- [Result] Inducing labour. London: National Institute for Health and Care Excellence (NICE); 2021 Nov 4. Available from http://www.ncbi.nlm.nih.gov/books/NBK579537/ PMID 35438865
- [Result] Kunt C, Kanat-Pektas M, Gungor AN, Kurt RK, Ozat M, Gulerman C, Gungor T, Mollamahmutoglu L. Randomized trial of vaginal prostaglandin E2 versus oxytocin for labor induction in term premature rupture of membranes. Taiwan J Obstet Gynecol. 2010 Mar;49(1):57-61. doi: 10.1016/S1028-4559(10)60010-1. PMID 20466294
- [Result] Gungorduk K, Asicioglu O, Besimoglu B, Gungorduk OC, Yildirm G, Ark C, Sahbaz A. Labor induction in term premature rupture of membranes: comparison between oxytocin and dinoprostone followed 6 hours later by oxytocin. Am J Obstet Gynecol. 2012 Jan;206(1):60.e1-8. doi: 10.1016/j.ajog.2011.07.035. Epub 2011 Jul 30. PMID 21924396
- [Result] Gulersen M, Zottola C, Li X, Krantz D, DiSturco M, Bornstein E. Chorioamnionitis after premature rupture of membranes in nulliparas undergoing labor induction: prostaglandin E2 vs. oxytocin. J Perinat Med. 2021 Jun 9;49(9):1058-1063. doi: 10.1515/jpm-2021-0094. Print 2021 Nov 25. PMID 34109770
- [Result] Mackeen AD, Durie DE, Lin M, Huls CK, Qureshey E, Paglia MJ, Sun H, Sciscione A. Foley Plus Oxytocin Compared With Oxytocin for Induction After Membrane Rupture: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jan;131(1):4-11. doi: 10.1097/AOG.0000000000002374. PMID 29215519
- [Result] Borovac-Pinheiro A, Inversetti A, Di Simone N, Barnea ER; FIGO Childbirth and Postpartum Hemorrhage Committee. FIGO good practice recommendations for induced or spontaneous labor at term: Prep-for-Labor triage to minimize risks and maximize favorable outcomes. Int J Gynaecol Obstet. 2023 Oct;163 Suppl 2:51-56. doi: 10.1002/ijgo.15114. PMID 37807591
- [Result] Middleton P, Shepherd E, Flenady V, McBain RD, Crowther CA. Planned early birth versus expectant management (waiting) for prelabour rupture of membranes at term (37 weeks or more). Cochrane Database Syst Rev. 2017 Jan 4;1(1):CD005302. doi: 10.1002/14651858.CD005302.pub3. PMID 28050900
- [Result] Dos Santos F, Drymiotou S, Antequera Martin A, Mol BW, Gale C, Devane D, Van't Hooft J, Johnson MJ, Hogg M, Thangaratinam S. Development of a core outcome set for trials on induction of labour: an international multistakeholder Delphi study. BJOG. 2018 Dec;125(13):1673-1680. doi: 10.1111/1471-0528.15397. Epub 2018 Sep 10. PMID 29981523
- See also: Royal Australian and New Zealand College of Obstetricians and Gynaecologists (RANZCOG). Term prelabour rupture of membranes (Term PROM). RANZCOG guideline [C-Obs 36]. Melbourne: RANZCOG; 2021 — https://ranzcog.edu.au/wp-content/uploads/Term-PROM.pdf